CLINICAL TRIAL: NCT06097013
Title: Science and Technology Innovation 2030
Brief Title: Study of Brain Function Evaluation System for Acute and Prolonged Disorders of Consciousness
Status: Enrolling by invitation | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Tianjin University (Other); Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021ZD0204300
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2023-08

CONDITIONS: Disorder of Consciousness
Keywords: Brain Function Test
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prolonged disorders of consciousness: Admission criteria for patients with prolonged disorders of consciousness Inclusion Criteria
  Interventions: Other: Routine clinical rehabilitation
- Acute disorders of consciousness: Admission criteria for patients with acute disorders of consciousness Inclusion Criteria
  Interventions: Other: Routine clinical rehabilitation

INTERVENTIONS:
Other: Routine clinical rehabilitation — Routine clinical rehabilitation

SUMMARY:
The research focuses on establishing a system for detecting loss of consciousness, developing clinical prognostic and awakening-related brain function testing criteria.

DETAILED DESCRIPTION:
A framework for the acquisition of neural features, feature selection and mechanism analysis of consciousness deficits in patients with acute and prolonged disorders of consciousness(DOC). Based on the multimodal data of three types of patients with DOC, the investigators established a comprehensive scientific collection of brain function features of acute and prolonged consciousness disorders; Revealed the key neural nodes and circuits of consciousness deficits, and elucidated the neural mechanisms of consciousness deficits in patients with prolonged consciousness disorders from EEG time-frequency-spatial features;

ELIGIBILITY:
Admission criteria for patients with prolonged disorders of consciousness

Inclusion Criteria:

1. Age 14-60 years;
2. In accordance with the diagnostic criteria of unresponsive arousal syndrome or minimally conscious state by international research;
3. Brain Trauma, stroke and hypoxic-ischemic encephalopathy lead to disturbance of consciousness;
4. right-handed；
5. The patient's family members signed the informed consent form;

Exclusion Criteria:

1. The history of mental illness and a history of hearing impairment;
2. Intracranial arterial clamp, pacemaker and other metal implants;
3. During the experiment, sedatives and other drugs that affect the excitability of the cortex;
4. The presence of uncontrolled seizures or involuntary movements;

Admission criteria for patients with acute disorders of consciousness

Inclusion Criteria:

(1)Age 14-60 years; (2）Meets diagnostic criteria for coma recognized in international studies； (3)the GCS score was less than 8; (4)Brain Trauma, stroke and hypoxic-ischemic encephalopathy lead to disturbance of consciousness; (5) right-handed； (6)The patient's family members signed the informed consent form;

Exclusion Criteria:

1. The history of mental illness and a history of hearing impairment;
2. Intracranial arterial clamp, pacemaker and other metal implants;
3. During the experiment, sedatives and other drugs that affect the excitability of the cortex;
4. The presence of uncontrolled seizures or involuntary movements; Admission criteria for patients with acute disorders of consciousness;
5. No spontaneous breathing;
6. Status Epilepticus;
7. Need emergency neurosurgical treatment can not cooperate with the examination;

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: prolonged disorders of consciousness and acute disorders of consciousness
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-04-13 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change from Coma recovery scale-revised | Within 24 hours of enrollment
  CRS-R scale includes 6 dimensions such as audiovisual, arousal level, verbal response, motor and communication, scoring 0 to 23, the higher the score the better the neurological function, and each score reflects the presence or absence of the evaluated person and the strength of consciousness
Change from the p300 in electroencephalogram | Assessment within 24 hours before, and 1 hour after TMS treatment
  Assessment the p300 in event related potential(ERP)
Change from resting-state in electroencephalogram | Assessment within 24 hours before, and 1 hour after TMS treatment
  Assessment the spectral power and coherence by in resting-state EEG
Change from TEP in electroencephalogram | Assessment within 24 hours before, and 1 hour after TMS treatment
  Assessment the TMS Evoked Potential(TEP)
Change from PCI in electroencephalogram | Assessment within 24 hours before, and 1 hour after TMS treatment
  Assessment the perturbational complexity index(PCI) in TMS-EEG

SECONDARY OUTCOMES:
Change from ROI in neuroimage techniques-PET | Assessment within 24 hours before ,and 1 hour after TMS treatment
  The distribution of 18F-FDG in the brain was analyzed according to the imaging situation, and the brain regions of interest (ROI) were outlined, and the uptake of 18F-deoxyglucose (FDG) in the patients was observed according to the brain ROI.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuan Wu hospitial, capical medical university, Beijing, China

IPD SHARING:
Plan to Share IPD: No